CLINICAL TRIAL: NCT03744143
Title: Comparison of Surgical Techniques for the Eradication of Deep Infiltrating Endometriosis of the Vagina: a Case-control Study
Brief Title: Surgical Eradication of Deep Infiltrating Endometriosis of the Vagina
Acronym: ENDO-VAG-r
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Principal Investigator, Mohamed Mabrouk, Principal investigator, IRCCS Azienda Ospedaliero-Universitaria di Bologna
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Endo-Vag
Record Dates: First submitted 2018-11-14; First posted 2018-11-16 (Actual); Last update posted 2019-04-02 (Actual); Status verified 2019-04

CONDITIONS: Endometriosis
Keywords: Vaginal endometriosis; Deep infiltrating endometriosis
MeSH Terms: conditions — Endometriosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (vaginal technique) (Other): Patients undergoing surgical removal of vaginal endometriotic nodule through vaginal technique
  Interventions: Procedure: Removal of vaginal endometriotic nodule
- Group B (laparoscopic technique) (Other): Patients undergoing surgical removal of vaginal endometriotic nodule through laparoscopic technique. Closure of the vagina with a transverse suture or a longitudinal suture.
  Interventions: Procedure: longitudinal suture; Procedure: transverse suture; Procedure: Removal of vaginal endometriotic nodule

INTERVENTIONS:
Procedure: longitudinal suture — Surgical eradication of deep infiltrating endometriosis of the vagina using laparoscopic technique, performing 4 transperitoneal abdominal accesses and trocars from 5 to 12 mm, and closure of the vagina with a longitudinal suture
  Arms: Group B (laparoscopic technique)
Procedure: transverse suture — Surgical eradication of deep infiltrating endometriosis of the vagina using laparoscopic technique, performing 4 transperitoneal abdominal accesses and trocars from 5 to 12 mm, and closure of the vagina with a transverse suture
  Arms: Group B (laparoscopic technique)
Procedure: Removal of vaginal endometriotic nodule — Surgical eradication of deep infiltrating endometriosis of the vagina using laparoscopic technique, performing 4 transperitoneal abdominal accesses and trocars from 5 to 12 mm, or vaginal technique, isolating the nodule through the vagina.

SUMMARY:
Multicentric retrospective study about the comparison of two different techniques of vaginal breach suturing after eradication surgery for deep infiltrating endometriosis and the surgical approaches (laparoscopic or vaginal) in terms of surgical, clinical and functional outcomes.

DETAILED DESCRIPTION:
Treatment of vaginal endometriosis can be successfully performed by vaginal or laparoscopic approach.

The results of the surgical treatment confirm its validity with regard to the reduction of dyspareunia in the short to medium term but show less efficacy in the long follow-up. The long-term impact of surgery on sexual function may be influenced by multiple factors, such as recurrence of symptomatic or anatomical disease, preservation of autonomic nerve fibers responsible for the arousal and genital sensitivity and residual vaginal length. These factors are potentially dependent on the surgical approach performed to treat vaginal endometriosis.

Particular importance as a surgical step assumes the closing phase of the vaginal defect that can be performed through a transverse or longitudinal suture. The longitudinal suture could guarantee, theoretically, a greater residual vaginal length and a better sexual function in the postoperative period than the vaginal closure by transversal suture, as demonstrated in previous studies about the suture techniques of vaginal cuff after hysterectomy.

Up to date, there are no studies comparing surgical, clinical and functional outcomes of the vaginal suture neither the two surgical approaches (laparoscopic or vaginal) for vaginal endometriosis eradication.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of vaginal endometriosis
* Women undergoing surgical removal with complete endometriotic lesions involving the vagina
* Informed consent for the processing of personal data for scientific purposes

Exclusion Criteria:

* History of previous or ongoing neoplastic pathology
* Patients committed to hysterectomy
* Previous vaginal surgery
* Not complete eradicating surgery
* Vaginism-vulvodynia
* Psychiatric disorders
* Genital prolapse
* Surgical menopause or spontaneous or pharmacological menopause

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 84 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2019-03-01 (Actual); Study Completion 2019-03-01 (Actual)

PRIMARY OUTCOMES:
Operative time | Intraoperative
  To compare the surgical techniques of vaginal endometriotic nodule removal considering the operative time

SECONDARY OUTCOMES:
Complication rate | Intraoperative
  Comparison of laparoscopic and vaginal approach concerning intraoperative complication rate in patients affected by vaginal endometriosis, using Clavien-Dindo Classification.
Evaluation of disease recurrence rate | Up to 6 months after surgery; from date of surgery until the date of first clinical or trans-vaginal/abdominal ultrasound documented recurrence, assessed up to 6 months
  Reappearance of vaginal nodule / rectum-vaginal septum in patients underwent different surgical techniques
Evaluation of dyspareunia recurrence rate | Up to 6 months after surgery
  Reappearance of dyspareunia in patients underwent different surgical techniques, assessed using a visual analog score, equal to or greater than 5
Complication rate | up to 30 days after surgery; from date of surgery until the date of first documented complication, assessed up to 30 days
  Comparison of laparoscopic and vaginal approach concerning complication rate in patients affected by vaginal endometriosis, using Clavien-Dindo Classification.

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - Gynecology and Physiopathology of Human Reproductive Unit, University of Bologna, S. Orsola-Malpighi Hospital, Bologna, BO
  - Policlinico Universitario Agostino Gemelli, Roma